CLINICAL TRIAL: NCT00823186
Title: Phase I Dose Escalation Study Of Weekly Paclitaxel and Cisplatin Followed by Radical Hysterectomy in FIGO IB2 and Bulky IIA Cervical Cancer
Brief Title: Dose-finding Study of Weekly Paclitaxel and Cisplatin in FIGO IB2 and Bulky IIA Cervical Cancer
Acronym: Chemothreapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Sinphar Pharmaceutical Co., Ltd (Other)
Responsible Party: Department of Obstetrics & Gynecology, Chang Gung Memorial Hospital, Kaohsiung
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-0365A3
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Cervical Cancer
Keywords: cervical carcinoma; neoadjuvant chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phyxol,cancer,intra vascular flow (Experimental): weekly cisplatin plus paclitaxel for 3 cycles as neoadjuvant chemotherapy (NAC) for FIGO IB2 and bulky IIA, squamous cell cervical cancer followed by radical hysterectomy and pelvic lymphedectomy
  Interventions: Drug: Phyxol(Paclitaxel)

INTERVENTIONS:
Drug: Phyxol(Paclitaxel) — Paclitaxel is 5ß,20-Epoxyl-1,2α,4,7,β 10 β,13 α-hexahydroxytax-11-en-9-one 4,10
  -diacetae 2-benzoate 13-ester with (2R,3S)-N-benzoyl-3-phenylisocerine

SUMMARY:
This phase I study is designed to establish an optimal dose of paclitaxel, under a fixed cisplatin dose at 40 mg/m2, delivered every week for three weeks, as neoadjuvant therapy before radical hysterectomy in bulky (FIGO IB2 or FIGO IIA with primary tumor dimension > 4 cm) squamous cell cervical cancer. This study will be conducted at all branches of Chang Gung Memorial Hospital.

The starting dose of paclitaxel is 50 mg/m2, and will be escalated by increments of 10 mg/m2 to a maximum dose of 80 mg/m2. The drugs will be administered sequentially (paclitaxel first, followed by cisplatin) within one day every week for three cycles.

A cohort of 3 patients, who are assessable for toxicity, is treated at each dose level. Each patient receives a fixed dose of paclitaxel and cisplatin, without modification. If none of the first 3 patients experiences a dose limiting toxicity (DLT, see definition below this paragraph), then escalation to the next dose level will proceed. If one patient develops a DLT, the cohort will be expanded to 6 patients. If no more than 1 of these 6 patients experiences a DLT, then escalation to the next dose level will proceed. The maximum tolerated dose (MTD) is the highest dose level at which no more than 1 of 6 patients experience a DLT. This dose level will be considered as the recommended dose for Phase II study. Although efficacy evaluation is not the main purpose of this study, a response rate of 60%, evaluated immediately before or at surgery, in all cases who have undergone 2 cycles of therapy is preset as a requirement for further phase II study using this regimen.The primary goal of NAC in cervical cancer is to improve the feasibility of surgical treatment, radical hysterectomy, without delaying the scheduled surgery or increasing the surgical risk or morbidity. Therefore, the definition of DLT for NAC is responded to this principle, in addition to the standard dose-limiting toxicity for phase I study.

DETAILED DESCRIPTION:
This is a multi-center, open-label, phase I study of paclitaxel and cisplatin as neoadjuvant therapy in patients with FIGO IB2 or bulky IIA, squamous cell cervical carcinoma of the uterine cervix.

The study is mainly for the dose-finding of paclitaxel, combining with a fixed cisplatinum dose, as neoadjuvant chemotherapy on a weekly basis. The optimal dose of paclitaxel is principally defined as the highest dose that allow at least 5/6 patients, after NAC, to undergo scheduled radical hysterectomy. A subsequent toxicity assessment to evaluate the impact of this neoadjuvant chemotherapy to the recovery of the following radical hysterectomy, and efficacy assessment is set as the second purpose of this study.

Primary Objectives:

* to establish an optimal dose of weekly cisplatin plus paclitaxel for 3 cycles as neoadjuvant chemotherapy (NAC) for FIGO IB2 and bulky IIA, squamous cell cervical cancer, followed by radical hysterectomy and pelvic lymphadenectomy

Secondary Objectives:

* to evaluate the toxicity of the study regimen and its impact to the radical hysterectomy after neoadjuvant chemotherapy
* to evaluate the overall tumor response to the neoadjuvant chemotherapy

An estimated of 8 to 21 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

women aged 35-70 years with all of the following criteria: untreated, histologically confirmed squamous cell carcinoma of the uterine cervix FIGO stage IB2 or bulky IIA, with tumor extension limited to within the upper one third of the vaginal wall. Bulky tumor is defined as (a) a visible cervical tumor with the largest diameter >4 cm or (b) a cervix expanded to > 4 cm as a result of tumor infiltration by pelvic examination and verified by magnetic resonance image (MRI), 3-dimensional (D) computed tomography (CT), or 3-D ultrasound study no suspicious lymph node metastasis as no enlarged lymph node or extrapelvic spread of cancer detected by MRI, or negative cytologic or histologic study of the suspicious node(s) (for those also participating PET-CT monitoring response trial, only abnormal FDG uptake in pelvic node(s) without proven nodal or extrapelvic metastasis are eligible)

Exclusion Criteria:

Histological or cytological documented pelvic lymph node or extrapelvic metastasis, concurrent or history of malignant tumor(s) other than treated nonmelanoma skin cancer had undergone surgical procedure other than cervical biopsy or had received cytotoxic procedure including chemotherapy, radiotherapy or treatment with biologic response modifier(s) for the cervical tumor participate in investigational treatment for the cervical cancer history of allergic reaction to platinum or paclitaxel uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements pregnant or breast feeding women, a urinary pregnancy test must be performed on all patients who are of child-bearing potential before entering the study and the result must be negative

-

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
to establish an optimal dose of weekly cisplatin plus paclitaxel for 3 cyclesas neoadjuvant chemotherapy (NAC) for FIGO IB2 and bulky IIA, squamous cell cervical cancer, followed by radical hysterectomy and pelvic lymphadenectomy | 18 months

SECONDARY OUTCOMES:
to evaluate the toxicity of the study regimen and its impact to the radical hysterectomy after neoadjuvant chemotherapy | 36 months
to evaluate the overall tumor response to the neoadjuvant chemotherapy | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: HAO LIN, MD, Principal Investigator — Chang Gung Memorial Hospital, Kaohsiung
Locations (3):
- Taiwan (3):
  - Chang Gung Memorial Hospital, Taoyuan District, Lin Kou
  - Chang Gung Memory Hpspital, Chiayi City
  - Taipei Chang Gung Memory Hospital, Taipei